CLINICAL TRIAL: NCT05237089
Title: Effects of Electroacupuncture on Weight Loss in Obese Patients With Prediabetes: a Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture on Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XSF20211230
Record Dates: First submitted 2021-12-28; First posted 2022-02-11 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Obesity
Keywords: Electroacupuncture; Obesity; Prediabetes; Sham acupuncture; Randomized Controlled Trial
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: All eligible participants will be randomly assigned into two group at a ratio of 1:1, the Electroacupuncture group and the Sham acupuncture group (the control group).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the acupuncturists in this study will know about the group assignment of patients. All other relevant parties will be blinded to the intervention. Participants will be informed that they will be randomly allocated to the electroacupuncture group or the superficial acupuncture group before study participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA group：Electroacupuncture+health education (Active Comparator): Acupuncture is the most popular adjuvant and alternative therapy in China, and it has been used to treat various diseases for thousands of years. Electroacupuncture is an innovation of traditional Chinese acupuncture, which improves the clinical effect by transmitting electrical pulses to the needles and then enhances the stimulation at the acupoints to receive better effects. Studies show that EA has been used as an alternative therapy for obesity in clinical practice.
  Interventions: Other: Electroacupuncture; Other: Health education
- Sham acupuncture group：shallow acupuncture+health education (Sham Comparator): Sham acupuncture method in this study is set as the superficial acupuncture manipulated at the same main acupoints with the thinner and shorter needles. The aim of the sham acupuncture is to eliminate the possible placebo effect of EA treatment.
  Interventions: Other: Sham acupuncture; Other: Health education

INTERVENTIONS:
Other: Electroacupuncture — Regular acupuncture will be applied at the main and the additional acupoints with 0.25mm*40mm or 0.30mm*75mm needles. The main acupoints include Shangwan (CV13), Zhongwan (CV12), Jianli (CV11), Xiawan (CV10), bilateral Quchi (LI11), Hegu (LI4), Liangmen (ST21), Tianshu (ST25), Daheng (SP15), Fujie (SP14), Shuidao (ST28), Zusanli (ST36), Fenglong (ST40), Wailing (ST26), Guilai (ST29). Additional acupoints include bilateral Shangjuxu (ST37) and Neiting (ST44), bilateral Yinlingquan (SP9) and Shuifen (CV9), Qihai (CV6) and Guanyuan (CV4). Acupuncturists will use all main acupoints and choose the combined acupoints based on the patients' patterns during each treatment session. The EA apparatus will be connected to the needles at the bilateral ST21, ST25, SP15, using continuous wave type, frequency at 3 Hz, and intensity of 4-5 mA based on the endurance of each patient. Needles will be retained for 30 minutes before removal.
  Arms: EA group：Electroacupuncture+health education
Other: Sham acupuncture — Patients will receive superficial acupuncture treatment at the same main acupoints as EA group with 0.22*0.25mm needles. The electroacupuncture apparatus will connected to the needles at the bilateral Liangmen (ST21), Tianshu (ST25), Daheng (SP15) without current output. Needles will be retained for 30 minutes before removal. The treatment will be given 3 times a week in week 1-12, 2 times a week in week 13-20, and once a week in week 21-24, totaling 56 sessions of real or sham acupuncture.
  Arms: Sham acupuncture group：shallow acupuncture+health education
Other: Health education — The health management brochure will be distributed to all patients in the trial after enrollment, and health education will be arranged online or offline at week 4, 8, 12, 16, 20 and 24 for about 60 minutes, including lifestyle, diet and physical activity. According to the specific situation of each patient, healthier individual lifestyle and behavior will be recommended to all patients, but there will be no strict restrictions on the diet or physical activity.

SUMMARY:
The investigators describe a protocol for a randomized controlled trial to find out the effect and safety of electroacupuncture on losing weight in obese patients with prediabetes.

DETAILED DESCRIPTION:
Obesity has emerged as a contributing factor in diabetes mellitus. In 2015, about 4 million deaths worldwide were directly related to high BMI, accounting for 7.1% of all deaths; among them, 41% died due to cardiovascular disease, followed by diabetes mellitus. China has become the country with the largest number of obese people and diabetic patients in the world. According to the clinical practice guidelines for medical care of obese patients announced by AACE and ACE, obese patients with prediabetes can effectively prevent the development of diabetes by lose 10% or more than of their body weight. Acupuncture is a widely recognized therapy to lose weight in clinical practice. But there are some doubts about the effectiveness of acupuncture versus sham acupuncture in treating obesity due to its lack of medical evidence.

This randomized placebo-controlled clinical trial is aimed to investigate the effect and safety of Electroacupuncture (EA) in obese patients with prediabetes. The investigators designed a protocol for a randomized controlled trial, in which 256 eligible patients will be randomly assigned to one of the two groups in a ratio of 1:1, the EA group (receiving EA treatment with health education) and the sham electroacupuncture (SA) group (receiving superficial acupuncture treatment with health education). A total of 56 sessions of interventions will be given for consecutive 24 weeks, followed by a 24-week follow-up period. Each session of EA or SA treatment will last for about 30 minutes. The primary outcome is the proportion of patients who lost 10% or more than of their body weight at week 24. The secondary outcomes include the change of patient's body weight and body mass index (BMI), results from the blood tests (FBG, 2hPG, HbA1c, HOMA-IR, LDL-C, HDL-C, TG and TC, ect.), the fat tissue size scanned by abdominal magnetic resonance imaging (MRI), data collected from the body composition analyzer, the and scores of the impact of weight on quality of life (IWQOL-Lite), Three Factor Eating Questionnaire - R21 (TFEQ-R21) and Food Cravings Questionnaire-Trait (FCQ-T). All adverse effects will be accessed by the Treatment Emergent Symptom Scale (TESS) from baseline to the follow-up period. The body weight and BMI will be calculated at baseline, week 8, week 16, week 24, week 32, week 40 and week 48, as well as the IWQOL-Lite, the TFEQ-R21 and the FCQ-T. Blood tests will be analyzed at baseline and week 24, as well as the body composition analyzer and the MRI scan. All patients will be provided with the same health education brochure to choose more beneficial personalized lifestyle during the 24-week intervention period.

All analyses will be performed on the intention-to-treat (ITT) population of participants who have at least one treatment. Missing data will be handled using the multiple imputation method, on the assumption that values at each time point follow a specific distribution calculated by the computer software R V.3.5. The primary analysis will be a comparison of the proportion of patients who losing 10% or more than of their body weight between the two groups at 24 weeks after inclusion (comparison of the primary endpoint). Linear mixed-effects models will be used for analyses with the use of the statistical software SPSS V.20.0. The t-test will be used to compare the measurement data between either two groups from the baseline to follow-up; the rank sum test will be used for ranked data while the Chi-squared test will be used to analyze categorical data. The significance level that will be used for statistical analysis with 2-tailed testing will be 2.5%. Data values will mainly be presented as Mean±SD.

The findings from this trial will help further explore the efficacy and safety of EA on losing weight for patients with obesity and prediabetes, as well as determine the differences between the EA and SA treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18-65;
2. Participant whose BMI is ≥24.0 kg/m2;
3. Participants whose HbA1c measurement of 5.7-6.4% both inclusive, or fasting plasma glucose measurement ≥ 6.1 mmol/liter and <7.0 mmol/liter, or 2-hour plasma glucose measurement post-challenge (oral glucose tolerance test) ≥7.8 mmol/liter and <11.1 mmol/liter;
4. Participants with stable weight within 3 months before the start of the trial, fluctuated within 4 kg;
5. Participants who voluntarily agree with the investigation and sign a written informed consent form for the clinical trial.

Exclusion Criteria:

1. Patients with secondary obesity caused by drugs or neuro-endocrine-metabolic disorders (such as hypothalamic disease and hypopituitarism);
2. Patients who have been diagnosed with type I or type II diabetes;
3. Patients who are taking medication which cause clinically significant weight gain or loss;
4. Patients whose Hamilton 17-item Depression Scale (HAMD-17) score >18 or have a history of other severe psychiatric disorders;
5. Patients with severe ulcer, abscess and skin infection at the local acupuncture area;
6. Patients with severe diseases of multiple organs, such as heart, brain, lungs, liver, kidneys, hematopoietic system or other serious diseases;
7. Participants who have joined in other clinical trials or studies within the past 1 month;
8. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Percentage of patients who lost 10% of their body weight | week 24
  We will calculate the proportion of people in each group who lost 10% or more of their baseline body weight at the end of the intervention period.

SECONDARY OUTCOMES:
Changes of body weight from baseline to week 48 | baseline, week 8, week 16, week 24, week 32, week 40 and week 48
  The change of body weight is an important factor of the development of diabetes. We will calculate the mean weight change in each group of patients during the intervention and follow-up period, compared with baseline data.
Changes of BMI from baseline to week 48 | baseline, week 8, week 16, week 24, week 32, week 40 and week 48
  BMI is a statistical index using a person's weight and height to provide an estimate of body fat in males and females of any age. It is calculated by taking a person's weight, in kilograms, divided by their height, in meters squared, or BMI = weight (kg)/ height2 (m2). BMI is used to define a person as underweight, normal weight, overweight, or obese by the National Institute of Health (NIH).
Change of blood glucose from baseline to week 24 | baseline, week 24
  It is the concentration of glucose in the blood, including fasting plasma glucose (FBG) which reflects function of islet β cell and 2 hour postprandial blood glucose (2hPG) which reflects the reserve function of islet β cell.
Change of HbA1c from baseline to week 24 | baseline, week 24
  HbA1c reflects the average blood glucose level of diabetic patients in the past 8-12 weeks. HbA1c≥5.5% indicates the presence of insulin resistance, and ≥6.5% indicates the occurrence of diabetes.
Change of insulin resistance index (HOMA-IR) from baseline to week 24 | baseline, week 24
  HOMA-IR is one of the most common formulas to reflect the intensity of insulin resistance. The higher index indicates the more serious insulin resistance. Insulin resistance index (HOMA-IR) = fasting insulin (FINS)*fasting plasma glucose (FPG)/22.5, HOMA-IR > 1 indicates the presence of insulin resistance.
Change of blood lipid from baseline to week 24 | baseline, week 24
  Blood lipid includes low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), triglyceride (TG), and total cholesterol (TC), which reflects the internal lipid metabolism of whole body.
Change of fat and muscle mass from baseline to week 24 | baseline, week 24
  The non-invasive body composition analyzer (Inbody 770) of the Inbody company can be used to measure high density body composition through bioelectrical impedance analysis, including body fat mass and skeletal muscle mass. The body fat mass reveals how much body fat makes up the weight, both surface level (subcutaneous) and internal (visceral). skeletal muscle mass is the muscle that can be grown and developed through exercise. And the muscle-fat analysis tells you whether you have a healthy balance of SMM and Body Fat Mass in respect to your weight.
Change of percentage body fat from baseline to week 24 | baseline, week 24
  The non-invasive body composition analyzer (Inbody 770) of the Inbody company can be used to measure high density body composition through bioelectrical impedance analysis, including percent body fat. Body fat percentage is a division of the participant's body fat mass by his/her total weight and a much better indicator of the risk of obesity than BMI.
Change of basal metabolic rate from baseline to week 24 | baseline, week 24
  The non-invasive body composition analyzer (Inbody 770) of the Inbody company can be used to measure high density body composition through bioelectrical impedance analysis, including the basal metabolic rate. BMR is the calories that one person needs for the basic essential functions. It allows the individual to work with the dietician to create a nutritional plan, which is key to reaching the body composition goals.
Change of fat tissue size from baseline to week 24 | baseline, week 24
  Abdominal magnetic resonance imaging (MRI) scan will be used to scan the upper abdomen and flat umbilical layer to quantitatively calculate abdominal fat size and the ratio of intra-abdominal and subcutaneous fat size.
Impact of weight on quality of life (IWQOL-Lite) | baseline, week 8,16, 24, 32, 40 and week 48
  It is a 31-item self-report questionnaire measuring the quality of life of obese patients (or those with type 2 diabetes). it consists of the following 5 dimensions: physical functioning, self-esteem, sexual life, public stress, and work included.
Three Factor Eating Questionnaire-R21(TFEQ-R21) | baseline, week 8,16, 24, 32, 40 and week 48
  TFEQ is one of the most widely used instruments to study different eating behaviors. It assesses three cognitive and behavioral domains of eating: cognitive restraint (6 items), uncontrolled eating (9 items) and emotional eating (6 items). It comprises 21 items in a four-point Likert scale for items 1-20 and on an eight-point numerical rating scale for item 21. Responses to each of the items are given a score between 1 and 4. Before calculating domain scores, items 1-16 were reverse coded and item 21 was recoded as follows: 1-2 scores as 1; 3-4 as 2; 5-6 as 3; 7-8 as 4.
Food Cravings Questionnaire-Trait (FCQ-T) | baseline, week 8,16, 24, 32, 40 and week 48
  It measures the frequency and intensity of food craving experiences in patients. The questionnaire has 39 items and response categories range from 1 = never to 6 = always. There are no inverted items. Responses to all items are summed up for a total score. Higher scores represent more frequent and intense food cravings.

OTHER OUTCOMES:
Adverse effects | from baseline to week 48
  Any adverse event (described as unfavourable or unintended signs, symptoms or diseases occurring during the trial) related to the intervention will be reported by patients and practitioners and accessed by the Treatment Emergent Symptom Scale (TESS) which is used as an associated indicator to mainly evaluate the safety of acupuncture treatment in this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shifen Xu, PhD, Study Director — Shanghai Municipal Hospital of Traditional Chinese Medicine
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data in this trial will be publicly available from the corresponding author upon reasonable request. All data and the protocol will be available after publication in peer-reviewed international journals for 3 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data and the protocol will be available after publication in peer-reviewed international journals for 3 years.
Access Criteria: The data in this trial will be publicly available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Li X, Lin J, Hu C, Liu B, Li F, Li J, Zeng X, Li S, Mi Y, Yin X, Xu S. Effect and safety of electroacupuncture on weight loss in obese patients with pre-diabetes: study protocol of a randomised controlled trial. BMJ Open. 2024 Mar 8;14(3):e075873. doi: 10.1136/bmjopen-2023-075873. PMID 38458786